CLINICAL TRIAL: NCT01998893
Title: Clinical Response in Patients With Relapsed Centroblastic Centrocytic Non-Hodgkin's Lymphoma After Treatment With Anti-CD20 Antibody IDEC C2B8 (MabThera)
Brief Title: A Study of MabThera/Rituxan (Rituximab) in Patients With Relapsed Centroblastic Centrocytic Non-Hodgkin's Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: M39004
Record Dates: First submitted 2013-11-25; First posted 2013-12-02 (Estimated); Results first posted 2014-11-04 (Estimated); Last update posted 2014-12-03 (Estimated); Status verified 2014-10

CONDITIONS: Non-Hodgkin's Lymphoma
MeSH Terms: conditions — Lymphoma, Non-Hodgkin | interventions — Rituximab

ARMS (1):
- MabThera/Rituxan (Experimental)
  Interventions: Drug: rituximab [MabThera/Rituxan]

INTERVENTIONS:
Drug: rituximab [MabThera/Rituxan] — 375 mg/m2 iv weekly for 4 weeks; for responders to first course of therapy a second course is possible after relapse

SUMMARY:
This study will evaluate the efficacy and safety of MabThera/Rituxan in patients with relapsed low-grade centroblastic centrocytic non-Hodgkin's lymphoma. Patients will receive once-weekly intravenous MabThera/Rituxan for 4 weeks; responding patients will be treated a second time in case of relapse (defined as progression after complete or partial response). The anticipated time on study treatment is <3 months.

ELIGIBILITY:
Inclusion Criteria:

* adult patients >= 18 years of age;
* centrocytic centroblastic non-Hodgkin's lymphoma stage III-IV;
* relapse after chemotherapy (with or without interferon maintenance therapy).

Exclusion Criteria:

* primary refractory lymphomas;
* more than 3 relapses of centroblastic centrocytic non-Hodgkin's lymphoma;
* clinically significant cardiac disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 1997-01; Primary Completion 2008-02 (Actual); Study Completion 2008-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (10):
- Germany (10):
  - Cologne
  - Erlangen
  - Göttingen
  - Grenzach-Wyhlen
  - Hanover
  - Homburg/saar
  - München
  - Münster
  - Stuttgart
  - Tübingen

RESULTS

PARTICIPANT FLOW:
Groups:
- Rituximab: Participants received rituximab, 375 milligrams per square meter (mg/m^2), intravenously (IV), over 4 hours, once per week for 4 weeks. Responders were eligible to receive a second course of treatment after relapse.
Period: Overall Study
Arm/Group | Rituximab
Started | 38
1st Treatment Cycle Completed Until PD | 30 (Progressive disease (PD))
2nd Treatment Cycle Started | 5
2nd Treatment Cycle Completed Until PD | 3
Completed | 21
Not Completed | 17
Not completed — Adverse Event | 2
Not completed — Death | 1
Not completed — Lost to Follow-up | 8
Not completed — Physician Decision | 2
Not completed — Protocol Violation | 2
Not completed — Withdrawal by Subject | 1
Not completed — Transformation to high-grade lymphoma | 1

BASELINE CHARACTERISTICS:
Population: Intent to treat (ITT) population included all participants with at least 1 application of study treatment.
Groups:
- Rituximab: Participants received rituximab, 375 mg/m^2, IV, over 4 hours, once per week for 4 weeks. Responders were eligible to receive a second course of treatment after relapse.
Arm/Group | Rituximab
Number analyzed (Participants) | 38
Age, Continuous [Median (Full Range); unit: years] | 55 [26 to 75]
Age, Customized [Number; unit: participants]
  Less Than or Equal to (≤) 18 Years | 0
  Between 18 and 65 Years | 32
  Greater Than or Equal to (≥) 65 Years | 6
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25
  Male | 13
Race (NIH/OMB) [Count of Participants; unit: Participants] — National Institutes of Health (NIH), Office of Management and Budget (OMB)
  Participants
    American Indian or Alaska Native | 0
    Asian | 0
    Native Hawaiian or Other Pacific Islander | 0
    Black or African American | 0
    White | 38
    More than one race | 0
    Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  Germany | 38
Ann Arbor stage [Number; unit: participants] — A staging system for lymphomas based on the location of the tumor and on systemic symptoms, ranging from stage I to stage IV.
  Stage III indicated that the cancer had spread to both sides of the diaphragm, including 1 organ or area near the lymph nodes or the spleen.
  Stage IV indicated diffuse or disseminated involvement of 1 or more extra-lymphatic organs, including any involvement of the liver, bone marrow, or nodular involvement of the lungs.
  participants
    Stage III | 5
    Stage IV | 33
Histological subtype [Number; unit: participants] — Histological subtype as confirmed by central pathologic review.
  participants
    Follicular or centroblastic/centrocytic lymphoma | 32
    Other | 6
B-Symptoms [Number; unit: participants] — B-Symptoms included high temperatures [greater than (>) 38 degrees Celsius (C)], night sweats, and unintentional weight loss >10 percent (%) over a period of 6 months or less.
  participants
    Present | 14
    Absent | 24
Bulky disease [Number; unit: participants] — Bulky disease was defined as at least 1 lesion ≥ 5 centimeters (cm) in diameter.
  participants
    Yes | 10
    No | 28
Bone marrow involvement [Number; unit: participants]
  Yes | 28
  No | 10
Liver involvement [Number; unit: participants]
  Yes | 6
  No | 32
Spleen involvement [Number; unit: participants]
  Yes | 16
  No | 21
  Missing | 1
Other extra-nodal lesions [Number; unit: participants]
  Yes | 8
  No | 30
Number of previous therapies [Number; unit: participants] — Number of previous therapies since diagnosis of lymphoma.
  participants
    1 previous therapy | 14
    2 previous therapies | 11
    3 previous therapies | 13

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With a Complete Remission (CR) or Partial Remission (PR)
Description: Percentage of participants with a CR, PR at the end of the first cycle of treatment (Week 4). CR was defined as the complete disappearance of all objective disease findings, including enlarged lymph nodes, hepatomegaly, and splenomegaly for at least 4 weeks, and a normalization of blood counts with granulocytes >1.500/ microliter (µL), hemoglobin (Hb) >12 grams per deciliter (g/dL), and platelets >100,000/µL. PR was defined as a less than (<) 50% regression of all measurable and evaluable lymphoma manifestations (sum of the products of the 2 largest diameters vertical to each other) for at least 4 weeks without the appearance of new manifestations, and normalization of blood counts.
Time Frame: Treatment start until progression of disease or last available follow-up. The median length of follow-up was 6.6 months (range: 0-97.8 months)
Population: ITT population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Rituximab
Number analyzed (Participants) | 38
percentage of participants | 39.5 [24.0 to 56.6]

2. Secondary Outcome: Number of Participants With a Clinical Response
Description: Clinical response was defined as the best response after the first 4 weeks of treatment cycle by the following categories: CR, PR, minor response (MR), stable disease (SD), and progressive disease (PD). CR was defined as the complete disappearance of all objective disease findings, including enlarged lymph nodes, hepatomegaly, and splenomegaly for at least 4 weeks, and a normalization of blood counts with granulocytes >1,500/μL, Hb >12 g/dL, and platelets >100,000/μL. PR was defined as <50% regression of all measurable and evaluable lymphoma manifestations (sum of the products of the 2 largest diameters vertical to each other) for at least 4 weeks without the appearance of new manifestations, and normalization of blood counts. MR was defined as tumor regression ≥25% and <50%. SD was defined as tumor regression <25%, no new manifestations, and progression ≤25%. PD was defined as no new lymphoma associated symptoms or an increase in the size of manifestations by more than 25%.
Time Frame: as for outcome 1
Population: ITT population
Measure: Number; unit: participants
Arm/Group | Rituximab
Number analyzed (Participants) | 38
participants
  CR | 9
  PR | 6
  MR | 3
  SD | 16
  PD | 2
  Missing | 2

3. Secondary Outcome: Time to Best Response
Description: The median time, in months, from start of the treatment (first application) until best response (PR or CR).
Time Frame: as for outcome 1
Population: ITT population; only participants with at least one application of study treatment within the first 4 weeks of treatment were included in the analysis.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Rituximab
Number analyzed (Participants) | 15
months | 1.9 [1.1 to 5.7]

4. Secondary Outcome: Duration of Remission
Description: Median time, in months, between the documentation of CR or PR and PD in clinical responders.
Time Frame: as for outcome 1
Population: Participants in the ITT population with CR or PR after the first treatment cycle.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Rituximab
Number analyzed (Participants) | 15
months | 12.7 [5.6 to 35.0]

5. Secondary Outcome: Time to Progression
Description: The median time, in months, from the start of treatment (first application) until detection of PD.
Time Frame: as for outcome 1
Population: ITT population
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Rituximab
Number analyzed (Participants) | 38
months | 6.6 [4.8 to 15.3]

6. Secondary Outcome: Overall Survival (OS)
Description: OS was defined as the time, in months, between enrollment into the study and death, due to any cause. Participants who were not reported as having died at the time of the analysis were censored using the date they were last known to be alive.
Time Frame: Enrollment into study until end of follow-up or death. The median length of follow-up was 6.6 months (range: 0-97.8 months)
Population: ITT population
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Rituximab
Number analyzed (Participants) | 38
months | 49.6 [15.3 to NA] — The statistical analysis system (SAS) could not compute the upper boundary of the confidence interval due to the large number of censored events.

7. Secondary Outcome: Number of Participants With a Clinical Response to Re-Treatment
Description: Clinical response was defined as the best response after the second 4 weeks of treatment cycle by the following categories: CR, PR, MR, SD, and PD. CR was defined as the complete disappearance of all objective disease findings, including enlarged lymph nodes, hepatomegaly, and splenomegaly for at least 4 weeks, and a normalization of blood counts with granulocytes >1,500/μL, Hb >12 g/dL, and platelets >100,000/μL. PR was defined as <50% regression of all measurable and evaluable lymphoma manifestations (sum of the products of the 2 largest diameters vertical to each other) for at least 4 weeks without the appearance of new manifestations, and normalization of blood counts. MR was defined as tumor regression ≥25% and <50%. SD was defined as tumor regression <25%, no new manifestations, and progression ≤25%. PD was defined as no new lymphoma associated symptoms or an increase in the size of manifestations by more than 25%.
Time Frame: First application in the second treatment cycle until progression of disease. The median length of follow-up was 4.6 months (range: 0.5-20.6 months).
Population: Participants in the ITT population who began a second cycle of treatment.
Measure: Number; unit: participants
Arm/Group | Rituximab
Number analyzed (Participants) | 5
participants
  CR | 1
  PR | 0
  MR | 0
  SD | 3
  PD | 0
  Missing | 1

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were reported from the beginning of study treatment until PD or last available follow-up in the first or the second treatment cycle. The median length of follow up was 6.7 months (range: 0-97.8 months).
Description: All participants who received at least 1 dose of study drug. AEs were collected according to the National Cancer Institute (NCI) Common Toxicity Criteria (CTC) Grading System revised on December 21st, 1994.
Arm/Group | Rituximab
Serious Adverse Events (participants affected / at risk) | 10/38
Other Adverse Events (participants affected / at risk) | 34/38
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Rituximab (N=38)
Allergy (Immune system disorders) | 1
Lymphocytes (Blood and lymphatic system disorders) | 2
Dysrhythmias (Cardiac disorders) | 1
Sinus tachycardia (Cardiac disorders) | 2
Lethargy (fatigue, malaise) (General disorders) | 1
Infection (Infections and infestations) | 1
Hypoglycemia (Metabolism and nutrition disorders) | 1
Shortness of breath (including wheezing) (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Rituximab (N=38)
Hemoglobine (Blood and lymphatic system disorders) | 3
Lymphocytes (Blood and lymphatic system disorders) | 5
Platelets (Blood and lymphatic system disorders) | 6
White blood count (Blood and lymphatic system disorders) | 3
Blood/bone marrow: other (not specified) (Blood and lymphatic system disorders) | 4
Dysrhythmias (Cardiac disorders) | 2
Sinus tachycardia (Cardiac disorders) | 2
Esophagitis/dysphagia/odonophagia (including recall reaction) (Gastrointestinal disorders) | 3
Nausea (Gastrointestinal disorders) | 5
Vomitting (Gastrointestinal disorders) | 3
Gastrointestinal: other (not specified) (Gastrointestinal disorders) | 3
Fever in absence of infection (including drug fever) (General disorders) | 14
Lethargy (fatigue, malaise) (General disorders) | 5
Myalgia (General disorders) | 2
Rigor/chills (grade 3 including cyanosis) (General disorders) | 12
Flue-like symptoms: other (not specified) (General disorders) | 4
Alkaline phosphatase (Hepatobiliary disorders) | 2
Bilirubin (Hepatobiliary disorders) | 2
Lactate dehydrogenase (LDH) (Hepatobiliary disorders) | 4
Alanine transaminase (ALT) (Hepatobiliary disorders) | 2
Hepatic: other (not specified) (Hepatobiliary disorders) | 3
Allergy (Immune system disorders) | 4
Infection (Infections and infestations) | 12
Coagulation: other (not specified) (Investigations) | 2
Hypokalemia (Metabolism and nutrition disorders) | 2
Metabolic: other (not specified) (Metabolism and nutrition disorders) | 6
Headache (Nervous system disorders) | 7
Sensory (Nervous system disorders) | 2
Neurologic: other (not specified) (Nervous system disorders) | 3
Genitourinary: other (not specifed) (Renal and urinary disorders) | 2
Shortness of breath (including wheezing) (Respiratory, thoracic and mediastinal disorders) | 2
Flushing (Skin and subcutaneous tissue disorders) | 2
Rash/itch (not due to allergy, including recall reaction) (Skin and subcutaneous tissue disorders) | 7
Skin: other (not specified) (Skin and subcutaneous tissue disorders) | 3
Edema (Vascular disorders) | 2
Hypotension (Vascular disorders) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.